CLINICAL TRIAL: NCT00697567
Title: Study in Healthy HSV Positive and HSV Negative Adults to Evaluate the Immunogenicity, Reactogenicity and Safety of GSK Biologicals' Herpes Simplex (gD) Candidate Vaccine With or Without Adjuvant
Brief Title: Evaluation of Immunogenicity, Reactogenicity and Safety of Herpes Simplex (gD) Candidate Vaccine With/Without Adjuvant
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Isabelle Harpigny, GSK
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 208141/002
Record Dates: First submitted 2008-06-12; First posted 2008-06-16 (Estimated); Last update posted 2008-06-16 (Estimated); Status verified 2008-06

CONDITIONS: Prophylaxis Herpes Simplex
Keywords: Herpes simplex; Herpes simplex vaccine
MeSH Terms: conditions — Herpes Simplex

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (4):
- Group A (Experimental): HSV seropositive subjects
  Interventions: Biological: Herpes simplex candidate vaccine GSK208141 - non-MPL-containing adjuvant
- Group B (Experimental): HSV seronegative subjects
  Interventions: Biological: Herpes simplex candidate vaccine GSK208141 - non-MPL-containing adjuvant
- Group C (Experimental): HSV seropositive subjects
  Interventions: Biological: Herpes simplex candidate vaccine GSK208141- MPL-containing adjuvant
- Group D (Experimental): HSV seronegative subjects
  Interventions: Biological: Herpes simplex candidate vaccine GSK208141- MPL-containing adjuvant

INTERVENTIONS:
Biological: Herpes simplex candidate vaccine GSK208141 - non-MPL-containing adjuvant — Intramuscular injection, 3 doses
  Arms: Group A; Group B
Biological: Herpes simplex candidate vaccine GSK208141- MPL-containing adjuvant — Intramuscular injection, 3 doses
  Arms: Group C; Group D

SUMMARY:
The purpose of the phase IIa study in healthy HSV seropositive and HSV seronegative adults is to evaluate the immunogenicity, reactogenicity and safety of herpes simplex (gD) candidate vaccine with or without adjuvant administered according to a 0, 1, 6 month schedule.

DETAILED DESCRIPTION:
At the time of conduct of this study, the sponsor GlaxoSmithKline was known by its former name SmithKline Beecham

ELIGIBILITY:
Inclusion Criteria:

* Between 18 and 40 years of age
* Written informed consent
* Female volunteers must be using contraceptive and should avoid becoming pregnant for the duration of this study.
* Good clinical condition as evidenced by history taking and physical examination

Exclusion Criteria:

* History of persistent hepatic, renal, cardiac or respiratory diseases.
* Clinical signs of acute illness at the time of entry into the study.
* Seropositive for antibodies against the human immunodeficiency virus (HIV).
* Pregnancy, lactation.
* Treatment with corticosteroids or immunomodulating drugs.
* Simultaneous participation in another clinical trial.
* Any previous history of allergy.
* Any concomitant vaccination or administration of immunoglobulin during the study period.
* Any abnormal laboratory value among the tests performed at screening

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 1992-09; Primary Completion 1997-12 (Actual); Study Completion 1997-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the immunogenicity of herpes simplex vaccine, with or without MPL, in healthy adult HSV seropositive and HSV seronegative volunteers | Days 0, 30, 60, 180 and 365 after vaccination
To evaluate the reactogenicity and safety of the MPL-containing and non-MPL-containing vaccine in healthy adult HSV seronegative and seropositive volunteers | Reactogenicity from day 0 to day 6 after vaccination. Safety from day 0 to day 365 after vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Clinical Trials Call Center, Ghent, Belgium